CLINICAL TRIAL: NCT03862677
Title: Determining Prognostic Immune Markers in Patients With Ovarian Cancer
Acronym: IMPrOVE
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, J.R. Kroep, Principal Investigator MD PhD, Leiden University Medical Center
Other Study IDs: NL66869.058.19
Record Dates: First submitted 2019-02-26; First posted 2019-03-05 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Epithelial ovarian cancer; Fallopian tube cancer; Primary peritoneal cancer; EOC; Immunity; IMPrOVE; Prognostic; Immune markers
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor material, ascites and blood samples before and/or during therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with (suspicion of) primary EOC
  Interventions: Other: No intervention
- Patients with recurrent EOC
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational study, no intervention

SUMMARY:
The IMPRoVE study is a prospective, non-interventional, explorative cohort study to determine prognostic immune markers in patients with epithelial ovarian cancer, fallopian tube cancer, and primary peritoneal cancer (EOC).

DETAILED DESCRIPTION:
Tumor material, ascites (if possible) and blood samples for immune monitoring will be collected from patients with primary and recurrent EOC undergoing surgery, chemotherapy and/or immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with (suspicion of) primary or recurrent EOC with an indication for surgery, chemotherapy and/or immunotherapy.
* Age ≥18 years.
* WHO performance status 0-2.
* Accessible for treatment and follow-up.
* Written informed consent.

Exclusion Criteria:

* Other active malignancy in past 5 years prior to entry into the study, except for treated non-melanoma skin cancer.
* Any known severe infection like HIV, hepatitis A, B and C.
* Receiving immune suppressive treatment.
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be carried out in patients with primary and recurrent EOC considered eligible for treatment with surgery, chemotherapy and/or immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Association between the mMDSC/DC ratio in PBMCs in patients with recurrent EOC before the start of treatment and OS | 5 years

SECONDARY OUTCOMES:
Association between the mMDSC/DC ratio in PBMCs in patients with recurrent EOC before the start of treatment and PFS | 5 years
Association between the mMDSC/DC ratio in PBMCs in patients with primary EOC before the start of treatment and OS | 5 years
Association between the mMDSC/DC ratio in PBMCs in patients with primary EOC before the start of treatment and PFS | 5 years
Interaction between the mMDSC/DC ratio in PBMCs and EOC groups on OS | 5 years
Interaction between the mMDSC/DC ratio in PBMCs and EOC groups on PFS | 5 years
Association between mMDSC/DC ratio in PBMCs measured at different time points in patients with primary EOC and OS | 5 years
Association between mMDSC/DC ratio in PBMCs measured at different time points in patients with recurrent EOC and OS | 5 years
Association between mMDSC/DC ratio in PBMCs measured at different time points in patients with primary EOC and PFS | 5 years
Association between mMDSC/DC ratio in PBMCs measured at different time points in patients with recurrent EOC and PFS | 5 years
Composition/counts of myeloid cells in PBMCs in patients with primary EOC before and during treatment and the association with OS | 5 years
Function of myeloid cells (assessed by functional suppression assay) in PBMCs in patients with primary EOC before and during treatment and the association with OS | 5 years
Composition/counts of myeloid cells in PBMCs in patients with recurrent EOC before and during treatment and the association with OS | 5 years
Function of myeloid cells (assessed by functional suppression assay) in PBMCs in patients with recurrent EOC before and during treatment and the association with OS | 5 years
Composition/counts of myeloid cells in PBMCs in patients with primary EOC before and during treatment and the association with PFS | 5 years
Function of myeloid cells (assessed by functional suppression assay) in PBMCs in patients with primary EOC before and during treatment and the association with PFS | 5 years
Composition/counts of myeloid cells in PBMCs in patients with recurrent EOC before and during treatment and the association with PFS | 5 years
Function of myeloid cells (assessed by functional suppression assay) in PBMCs in patients with recurrent EOC before and during treatment and the association with PFS | 5 years
Influence of the mMDSC/DC ratio and separate immune cell populations on the tumor specific and general immune response (assessed by mixed lymphocyte reaction, functional suppression assay and lymphocyte stimulation test) | 5 years
Determined, optimized and validated optimal cut-off point for the macrophage/DC ratio and the mMDSC/DC ratio in PBMCs in patients with primary EOC for the different chemotherapeutic and immunotherapeutic treatment modalities | 5 years
Determined, optimized and validated optimal cut-off point for the macrophage/DC ratio and the mMDSC/DC ratio in PBMCs in patients with recurrent EOC for the different chemotherapeutic and immunotherapeutic treatment modalities | 5 years
Immune contexture of primary tumors by determination of the intratumoral immune subset numbers in fresh and archived tumor material and the association with OS | 5 years
Immune contexture of recurrent tumors by determination of the intratumoral immune subset numbers in fresh and archived tumor material and the association with OS | 5 years
Immune contexture of primary tumors by determination of the intratumoral immune subset numbers in fresh and archived tumor material and the association with PFS | 5 years
Immune contexture of recurrent tumors by determination of the intratumoral immune subset numbers in fresh and archived tumor material and the association with PFS | 5 years
Immune contexture of ascites by determination of the immune subset numbers in ascites fluid of patients with primary EOC and the association with OS | 5 years
Immune contexture of ascites by determination of the immune subset numbers in ascites fluid of patients with recurrent EOC and the association with OS | 5 years
Immune contexture of ascites by determination of the immune subset numbers in ascites fluid of patients with primary EOC and the association with PFS | 5 years
Immune contexture of ascites by determination of the immune subset numbers in ascites fluid of patients with recurrent EOC and the association with PFS | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Judith R Kroep, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided